CLINICAL TRIAL: NCT01427023
Title: Prospective Collection of Female First-catch Urine, Vaginal Swab, Endocervical Swab, and Cervical Specimens for Testing With the APTIMA Trichomonas Vaginalis Assay
Brief Title: Female Urine, Vaginal & Endocervical Swab & Cervical Specimen Collections for APTIMA Trichomonas Vaginalis Assay Testing
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: ATVPS-US11-001
Record Dates: First submitted 2011-08-26; First posted 2011-09-01 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Trichomonas Vaginalis
Keywords: APTIMA Trichomonas vaginalis Assay; APTIMA; trichomonas; trichomonas vaginalis
MeSH Terms: conditions — Trichomonas Infections | interventions — Biological Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine specimen, vaginal swab specimen, endocervical swab specimen and PreservCyt specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APTIMA Trichomonas vaginalis (ATV) Assay — APTIMA Trichomonas vaginalis (ATV) Assay

SUMMARY:
The objective of this study is to obtain female first-catch urine, vaginal swab, endocervical swab, and cervical specimens collected in PreservCyt Solution ("PreservCyt Specimens") for testing with the APTIMA Trichomonas vaginalis (ATV) Assay.

These specimens will be used to demonstrate assay performance on the PANTHER System is comparable to performance on the TIGRIS System.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be female and attend a participating clinic
* Subject must be at least 14 years of age at the time of enrollment and is currently sexually active (has had vaginal intercourse within the past 12 months)
* The subject and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented consent of her parent or legal guardian, unless the site has an institutional review board (IRB)- approved waiver for parental consent for minors)
* In addition, the subject must meet at least one of the following criteria:

  * Subject must demonstrate symptoms consistent with a suspected STD such as vaginal odor, vaginal discharge, vaginal/vulvar itching or irritation, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort
  * Subject must be asymptomatic and known to be partners with, or a contact of, a person with a confirmed or suspected STD(s)
  * Subject must be asymptomatic and undergoing screening evaluation for possible STDs
  * Subject must be undergoing Pap screening

Exclusion Criteria:

* Subject took antibiotic medications within the last 14 days
* Subject already participated in the study
* Subject has a history of illness that the principal investigator (PI) or designee considers could interfere with or affect the conduct, results, and/or completion of the clinical trial
* Subject has a history of illness that the PI or designee considers could create an unacceptable risk to the subject if enrolled

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women attending participating US OB/GYN, family planning, or STD clinics will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Positive Percent Agreement Using the TIGRIS Instrument as a Reference. | approximately one year
  Positive Percent Agreement Using the TIGRIS Instrument as a Reference.
Negative Percent Agreement Using the TIGRIS Instrument as a Reference. | approximately one year
  Negative Percent Agreement Using the TIGRIS Instrument as a Reference.

SECONDARY OUTCOMES:
Positivity Rate | approximately one year
  Positivity Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Wishard Hospital - Indiana University School of Medicine, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - New England Center for Clinical Research, Fall River, Massachusetts
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Geneuity Clinical Research Services, Maryville, Tennessee
  - Planned Parenthood Gulf Coast, Houston, Texas